CLINICAL TRIAL: NCT06104683
Title: A Phase 2, Randomized Study of Pirtobrutinib Versus Placebo in Patients With Relapsing Multiple Sclerosis
Brief Title: A Study of Pirtobrutinib (LY3527727 [LOXO-305]) Versus Placebo in Participants With Relapsing Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision: The trial has been withdrawn with no plans to continue development.
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18690; J2N-MC-KLAA (Other: Eli Lilly and Company); 2022-502376-24-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-10-24; First posted 2023-10-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Relapsing Multiple Sclerosis; Multiple Sclerosis
Keywords: Relapsing Forms Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — pirtobrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pirtobrutinib Dose 1 (Experimental): Participants will receive pirtobrutinib orally.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib Dose 2 (Experimental): Participants will receive pirtobrutinib orally.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib Dose 3 (Experimental): Participants will receive pirtobrutinib orally.
  Interventions: Drug: Pirtobrutinib
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Pirtobrutinib — Administered orally
  Other Names: LY3527727
  Arms: Pirtobrutinib Dose 1; Pirtobrutinib Dose 2; Pirtobrutinib Dose 3

SUMMARY:
The main purpose of this study is to assess efficacy and safety of pirtobrutinib in participants with relapsing multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been diagnosed with relapsing MS
* Participants must have one of the following

  1. at least 1 documented relapse within the previous year, or
  2. at least 2 documented relapse within the previous 2 years, or
  3. at least 1 active Gd-enhancing brain lesion on an MRI scan in the past 6 months prior to screening.

Exclusion Criteria:

* Have had a diagnosis of primary progressive MS
* Have a history of another clinically significant neurological disease
* Had a relapse of MS within 30 days prior to randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
New T1 Gadolinium (Gd)-enhancing Lesions on Brain Magnetic Resonance Imaging (MRI) Per Scan | Week 8 and Week 12
Number of New and/or Enlarging T2 Lesions | Week 12

SECONDARY OUTCOMES:
Total Number of T1 Gd-Enhancing Lesions Per Scan | Week 8 and Week 12
Total Number of Gd-Enhancing Lesions Per Scan | Week 8 and Week 12
Pharmacokinetics (PK): Plasma Concentration of Pirtobrutinib | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (3):
  - University of South Florida, Tampa, Florida
  - Clinical Trial Network, Houston, Texas
  - Swedish Medical Center-501 E Hampden Ave, Seattle, Washington
- Caribbean Center For Clinical Research Inc, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/